CLINICAL TRIAL: NCT06531525
Title: A Multicenter, Open-label, Randomized, Controlled, Phase 2 Trial Evaluating Whether Low Molecular Heparin Could Improve Pregnancy Outcomes With Protein S Deficiency
Brief Title: Effect of Low Molecular Heparin on Pregnancy Outcome With Protein S Deficiency
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other); China-Japan Friendship Hospital (Other); Sichuan Academy of Medical Sciences (Other); Xiangya Hospital of Central South University (Other); Chinese PLA General Hospital (Other); Beijing Friendship Hospital (Other); Beijing Chuiyangliu Hospital (Other Government)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PKU-PS-01
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Related; Protein S Deficiency
Keywords: Protein S Deficiency; pregnancy; therapy
MeSH Terms: conditions — Protein S Deficiency | interventions — Enoxaparin; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The combination group (Experimental): Subjects randomized to the combination group will receive daily injections of enoxaparin at a dose of 4000 IU and aspirin 75mg per day orally until delivery.
  Interventions: Drug: Enoxaparin; Drug: Aspirin
- The Aspirin group (Active Comparator): Aspirin will be given at a dose of 75mg, orally, each day until delivery.
  Interventions: Drug: Aspirin
- No intervention (No Intervention): No intervention
- All groups (Other): Participants in all groups will receive daily injections of enoxaparin at a dose of 4000 IU within 6 weeks at postpartum.
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin 4000 IU/day by subcutaneous injection at the time of randomization and continued until delivery. Dose adjustments were made throughout the study based on symptoms such as bleeding and thrombosis.
  Other Names: lovenox; clexane
  Arms: The combination group
Drug: Aspirin — Aspirin 75mg, orally, once daily at the time of randomization and continued until delivery. Dose adjustments were made throughout the study based on symptoms such as bleeding and thrombosis.
  Other Names: ASA
  Arms: The Aspirin group; The combination group
Drug: Enoxaparin — Participants in all groups will receive daily injections of enoxaparin at a dose of 4000 IU within 6 weeks at postpartum.
  Other Names: lovenox; clexane
  Arms: All groups

SUMMARY:
To evaluate whether low molecular heparin could improve pregnancy outcomes in pregnancies with protein S deficiency.

DETAILED DESCRIPTION:
This is a parallel-group, multicenter, randomized controlled trial of 48 pregnancies with protein S deficiency in China. Patients are randomized into three groups to receive enoxaparin combined with aspirin, aspirin alone and no intervention. The primary outcome measure is livebirth rate.

ELIGIBILITY:
Inclusion Criteria:

1. Plasma activity levels of PS when not pregnant are below the lower limits of the adult reference values (generally about 60-70% for PS) without the use of warfarin. Or, free protein S antigen levels in the second and third trimesters are less than 30% and less than 24%, respectively
2. Pregnant women who delivered from Aug 1st, 2024 to Oct 15th, 2027
3. One or more family members exhibiting the same symptoms as the patient
4. Past history of early onset thrombosis (age 50 or below)
5. Repeated recurrence of thrombosis
6. Thromboses in unusual sites
7. New onset of thrombosis during current pregnancy or after delivery
8. Patients with diagnosis confirmed by gene analysis Inclusion criteria 1 and 2 must always be met regardless of items of 3-8.
9. Written informed consent

Exclusion Criteria:

1. Thrombophilia other than Protein S deficiency
2. Antiphospholipid syndrome, systemic lupus erythematosus, platelet abnormalities, vascular disorders, blood flow obstruction, paroxysmal nocturnal hemoglobinuria, malignant tumor and other conditions that tend to cause thrombosis
3. Allergy/hypersensitivity to enoxaparin or aspirin
4. Heparin-associated thrombocytopenia or thrombocytopenia (platelet count<75 × 10^9/L)
5. Organ lesions at risk for bleeding such as acute stomach/bowel ulcers, cerebral hemorrhage, cerebral aneurysm
6. uncontrolled hypertension or Severe hypertension (Systolic Blood Pressure >200mmhg and/or Diastolic Blood Pressure >120mmHg)
7. Severe hepatic failure (INR >1.8)
8. Serum creatinine greater than 80 umol/L (1.3mg/dl) and an abnormal 24 hour urine creatine clearance (<30ml/min)
9. Abnormal uterine cavity on hysterosalpingogram/hysteroscopy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of livebirth | From date of randomization until delivery, assessed up to 42 months
  Incidents of livebirth

SECONDARY OUTCOMES:
Parameters of maternal coagulation-related indicators | From the start of study treatment to 6 weeks post-partum
  D-Dimer in ng/ml, Protein S activity in %
Parameters to assess the safety of low molecular heparin | From the start of study treatment to 6 weeks post-partum
  Maternal platelet count in 10^9/L, Number of haemorrhagic events, Number of cases of skin reactions at injection site
Other incidents of adverse pregnancy outcomes | up to 37 weeks
  early miscarriage (until 12 weeks of gestation), late miscarriage (12-28 weeks of gestation), premature livebirths (28-37 weeks of gestation)
Neonatal Data | after the delivery (an expected average of one month)
  Neonatal weight in grams, Neonatal length in centimetres, Apgar 1-minute, 5-minute, 10-minute scores in scores, Number of neonatal complications
Incidents of placental insufficiency | up to 6 weeks post-partum
  Incidents of pre-eclampsia, intrauterine growth retardation, placental abruption, and intrauterine foetal death, etc.
Incidents of thrombosis/thromboembolism | From the start of study treatment to 6 weeks post-partum
  thrombosis/thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, Professor, Principal Investigator — Peking University Insititute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing/Beijing, China